CLINICAL TRIAL: NCT07017972
Title: Multicenter Data Collection and Simulated-Use Assessment for CHLOE
Brief Title: Data Collection and Professional Simulated Use Study to Develop an Embryo Quality Artificial Intelligence (AI) Model
Status: Recruiting | Type: Observational
Sponsor: Fairtility (Industry)
Responsible Party: Sponsor
Other Study IDs: FRT-25-01
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: AI evaluation of embryos — AI evaluation of embryos inside a time-lapse incubator.

SUMMARY:
This protocol supports the reliable development and improvement of Artificial Intelligence (AI)-based applications by enabling training, verification, and validation using high-quality real clinical data. It also aims to enhance machine learning in developmental-use AI software.

In addition, the professional user simulated use will ensure correct and easy use of the AI applications.

DETAILED DESCRIPTION:
This data collection protocol aims to allow the reliable and robust development (training, verification, and validations) of Artificial Intelligence (AI) technology-based applications as well as improving the machine learning stage of released devices/applications - an AI - based software, for developmental use only, through inspection of large body of high quality real clinical data. Another important element in the design of the application is the user interface. It is thus important to run simulated use assessments to ensure correct and easy use of the AI application by professional users.

ELIGIBILITY:
Inclusion Criteria:

1. Images and data of eggs or embryos available from egg retrievals by women undergoing standard egg-freezing or In vitro fertilization (IVF) treatments, using their own eggs or donor eggs.
2. Women at least 18 years of age.
3. Embryos or eggs cultured in a time-lapse incubator connected to the AI Embryo Viewer.

Exclusion Criteria:

* Women with no available own or donor eggs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women undergoing In vitro fertilization (IVF) treatment
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) will be quantified using logistic regression to assess EQ Score's prediction of utilization. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Wiemer, PhD, Study Chair — Fairtility
Locations (1):
- New England Fertility Institute, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided